CLINICAL TRIAL: NCT00179322
Title: Effects of Sleep Deprivation and Recovery Sleep on Speech, Language and Other Higher Cognitive Functions: A Combined EEG-fMRI Study
Brief Title: Effects of Sleep Deprivation and Recovery on Cognitive Functions
Status: Completed | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050238; 05-DC-0238
Record Dates: First submitted 2005-09-15; First posted 2005-09-15 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-09-30

CONDITIONS: Sleep Deprivation
Keywords: Sleep Architecture; Sleep Measures; Speech Articulation; Cerebral Perfusion; Neuroimaging; Healthy Volunteer; HV
MeSH Terms: conditions — Sleep Deprivation

SUMMARY:
This study will measure brain activity in individuals performing language tasks while in various states of alertness to learn more about how the central nervous system is affected by impairments such as sleepiness.

Healthy normal volunteers between 20 and 40 years of age may be eligible for this study. Candidates must be non-smokers, right-handed, speak English fluently and have at least 12 years of education. They are screened with a medical history, physical examination, hearing and speech evaluation, computer task training, blood and urine tests and a late-night functional magnetic resonance imaging (fMRI) scan (see description below). Before screening and again before participating in the study, candidates wear an actigraph (a wristwatch-like device that records motion) for 7 days to provide a measure of their sleep-wake patterns.

Participants undergo the following tests and procedures:

* Extended wakefulness: Subjects are kept awake longer than is normal for them in their everyday life to be able to examine the brain under conditions of sleepiness. They are engaged in activities with the research staff during this waking time.
* Functional magnetic resonance imaging: Subjects undergo five separate fMRI scans-one during screening and four others during the main part of the study. fMRI uses a magnetic field and radio waves to produce images of the brain. The subject lies on a table that is moved into the scanner (a narrow cylinder), wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. Brain scans are taken at rest and while the subject performs tasks, which include pressing a button upon seeing certain shapes and performing various language tasks, such as saying memorized or new words, listening to narratives, and describing everyday procedures.
* Neurological, speech-language, and neuropsychological testing: Before the fMRI exams and during the period of extended wakefulness, subjects complete a series of tests that measure speech, language, memory and visual skills. Portions of the tests may be video- or autiotaped.
* Interviews and questionnaires: Participants are interviewed about their handedness, sleep history, and presence of medical or neurological symptoms.
* Electrophysiological studies: Subjects have an electroencephalograph (EEG) to measure the electrical activity of the brain and surface electromyography (EMG) to measure movements of muscles involved in moving and speaking. For the EEG, electrodes (small metal disks) are attached to the surface of the scalp or to a cap placed over the head. For the EMG, electrodes are attached to the skin of the face and neck by plastic or paper tape.

DETAILED DESCRIPTION:
Objectives of this protocol are to examine fMRI data taken concurrently with speech, language, and decision making tasks under conditions of both alertness and sleep deprivation, comparing fMRI-defined neural activation across states and behavioral performance, assessing changes in brain function with sleep deprivation. An additional objective is to develop an fMRI signal based sleep scoring system. Subjects will be 45 normal healthy volunteers, age 20-40, who meet criteria both for safe participation in an fMRI environment and for suitability for research on normal human sleep. To examine speech and language processing and also to examine depth of sleep, we will use a within-subjects free behavior design in which we search for patterns in the arterial spin labeled (ASL) or the blood oxygen dependent (BOLD) signal in fMRI data recorded while subjects say rehearsed word sets, describe or listen to novel procedures, or transition from wake to sleep. To gauge subjects' speech and language, we will record, concurrently with fMRI, their voice for analysis in conditions of both alertness and sleep deprivation. To examine decision making, we will compare the fMRI signal during response execution and inhibition across conditions of alertness and sleep deprivation. To gauge subjects' depth of sleep during fMRI, we will use both physiological (e.g., EEG) and behavioral measures (e.g., latency and quality of rehearsed verbal response to external stimuli presented during sleep). For speech, language processing, and depth of sleep, key measures will include fundamental frequency, speaking rate, voice onset, word production, and linguistic variables (phonological, syntactic, and pragmatic) derived from recorded transcripts. For decision making, the key measure will be subjects' errors and latencies in responding to cues to make or refrain from making a prescribed action. The fMRI data corresponding to these behavioral data are expected to show systematic changes in neural activation patterns that parallel behavioral changes with sleep deprivation.

ELIGIBILITY:
* INCLUSION CRITERIA:

Normal healthy volunteers in this protocol should be fluent English speaking and have at least 12 years of education.

Subjects should also be right-handed.

EXCLUSION CRITERIA:

People who are not native speakers of English or are left handed will be excluded from this study.

Given the nature of the stimuli presentation (i.e., projected visual images and speakers carrying voice), anyone with noncorrectable vision impairments, hearing loss, or known risk for hearing loss will be excluded. Normal hearing is defined as hearing thresholds of 25dB HL or less for the octave frequencies 250 - 8000 Hz and intact crossed acoustic reflex in both ears.

The dual focus of this research on sleep deprivation and fMRI yields additional sets of exclusion criteria for both fMRI safety and normal sleep/wake patterns. Given the dimensions of the fMRI and the exam table, anyone whose body size or shape cannot be accommodated in the fMRI with a projected image remaining continuously visible will be excluded.

Women who are pregnant will be excluded from this protocol.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2005-09-10; Study Completion 2016-09-30

CONTACTS AND LOCATIONS:
Overall Officials: Allen R Braun, M.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] ASERINSKY E, KLEITMAN N. Regularly occurring periods of eye motility, and concomitant phenomena, during sleep. Science. 1953 Sep 4;118(3062):273-4. doi: 10.1126/science.118.3062.273. No abstract available. PMID 13089671
- [Background] Bechara A, Damasio AR, Damasio H, Anderson SW. Insensitivity to future consequences following damage to human prefrontal cortex. Cognition. 1994 Apr-Jun;50(1-3):7-15. doi: 10.1016/0010-0277(94)90018-3. PMID 8039375
- [Background] Bechara A, Tranel D, Damasio H, Damasio AR. Failure to respond autonomically to anticipated future outcomes following damage to prefrontal cortex. Cereb Cortex. 1996 Mar-Apr;6(2):215-25. doi: 10.1093/cercor/6.2.215. PMID 8670652